CLINICAL TRIAL: NCT05338177
Title: Pilot Trial on Immunosuppression Modulation in Kidney Transplant Recipients Without SARS-CoV-2 Spike Protein Antibodies Following Full Vaccination
Brief Title: Pilot Trial on Immunosuppression Modulation to Increase SARS-CoV-2 Vaccine Response in Kidney Transplant Recipients
Acronym: BOOST_TX_SubA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Roman Reindl-Schwaighofe, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BOOST_TX_SubA
Record Dates: First submitted 2022-04-08; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunosuppression reduction (Experimental): Participants stop mycophenolate or azathioprine for two weeks peri-vaccination. Treatment is stopped on week before vaccination and only restarted one week after vaccination
  Interventions: Other: Immunosuppression reduction
- No immunosuppression reduction (Active Comparator): no alterations to immunosuppression
  Interventions: Other: No immunosuppression reduction

INTERVENTIONS:
Other: Immunosuppression reduction — participants stop mycophenolate or azathioprine one week before additional vaccine dose. Overall medication is stopped for two weeks.
  Arms: Immunosuppression reduction
Other: No immunosuppression reduction — participants do not alter immunosuppresion
  Arms: No immunosuppression reduction

SUMMARY:
Mycophenolate has been identified as risk factor for non-response to SARS-CoV-2 vaccination in kidney transplant recipients. Safety and efficacy of temporarily stopping of mycophenolate (or azathioprine) to increase vaccine response has not been established.

This is a non-randomized, controlled pilot study including up to 40 kidney transplant recipients not responding to at least three previous SARS-CoV-2 vaccine doses. Mycophenolate or azathioprine will be stopped for two weeks peri-vaccination starting one week before vaccination until one week after vaccination. Allocation to mycophenoalte or azathioprine discontinuation arm will be based on an overall risk assessment by the transplant physician and patient preference. Patients not stopping mycophenolate or azathioprine will serve as control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received a kidney transplantation
* > 18 years of age
* No SARS-CoV-2 spike protein antibodies four weeks after at least three previous vaccine doses
* Maintenance immunosuppression with mycophenolate or azathioprine

Exclusion Criteria:

* acute illness with fever
* Prior documented infection with SARS-CoV-2
* triple anticoagulation therapy
* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s)
* Subject has known sensitivity or intolerance to any of the products to be administered for the purpose of this study
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with the study procedures
* Subject is pregnant or breast feeding
* SARS-CoV-2 spike protein antibodies four weeks after the 3rd last vaccination > 0.8 BAU/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-11-14 (Estimated)

PRIMARY OUTCOMES:
Seroconversion at 4 weeks | 4 weeks
  Number of patients developing SARS-CoV-2 antibodies at 4 weeks after vaccination

SECONDARY OUTCOMES:
Seroconversion at 7 days | 7 days
  Number of patients developing SARS-CoV-2 antibodies at 7 days after vaccination
Antibody levels at 4 weeks | 4 weeks
  SARS-CoV-2 antibody levels at 4 weeks after vaccination
Donor specific antibodies | 4 weeks
  Donor specific antibodies at 4 weeks after mycophenolate / azathioprine pausing
Donor-derived cell free DNA | 4 weeks
  Donor-derived at 4 weeks after mycophenolate / azathioprine pausing
Creatinine levels | 4 weeks
  Creatinine levels at 4 weeks after mycophenolate / azathioprine pausing

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No